CLINICAL TRIAL: NCT05269134
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Safety and Efficacy of APT Phage Bank Phage Therapy Versus Placebo in Conjunction With Debridement, Antibiotics, and Implant Retention (DAIR) in Subjects With Chronic Prosthetic Joint Infection (PJI)
Brief Title: Bacteriophage Therapy in Patients With Prosthetic Joint Infections (PJI)
Acronym: ACTIVE2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Adaptive Phage Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APT.PJI.006
Record Dates: First submitted 2022-02-25; First posted 2022-03-07 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-10

CONDITIONS: Prosthetic Joint Infection
Keywords: Prosthetic; Joint; Knee; Hip; Phage; Bacteriophage; Prosthetic Joint; DAIR

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DAIR + Phage Treatment + Antibiotics (Experimental): Phage therapy will be administered in conjunction with antibiotic treatment.
  Interventions: Drug: Bacteriophage
- DAIR + Placebo + Antibiotics (Placebo Comparator): Placebo will be administered in conjunction with antibiotic treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bacteriophage — Phage Therapy
  Arms: DAIR + Phage Treatment + Antibiotics
Drug: Placebo — Placebo
  Arms: DAIR + Placebo + Antibiotics

SUMMARY:
This is a study designed to evaluate bacteriophage therapy in patients with chronic prosthetic joint infections.

DETAILED DESCRIPTION:
This is a study designed to evaluate bacteriophage therapy in patients with chronic prosthetic joint infections of the hip or knee caused by at least 1 of the following organisms: Staphylococcus aureus, Staphylococcus epidermidis, Staphylococcus lugdunensis, Streptococcus spp., Enterococcus faecium, Enterococcus faecalis, Escherichia coli, Pseudomonas aeruginosa, or Klebsiella pneumoniae.

This study will compare the safety and efficacy of DAIR procedure + Phage Therapy + Antibiotics versus DAIR procedure + Placebo + Antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥18 years of age
* Recurrent PJI of the knee or hip
* Female patients of childbearing potential who agree to use contraception.
* Confirmed phage match
* No anticipated need for long-term antibiotics

Exclusion Criteria:

* Soft tissue defect requiring reconstruction
* Hardware misalignment
* Additional orthopedic hardware in connection with the infected prosthesis
* Active infection (other than PJI) requiring long term IV antibiotics
* Unable to tolerate SAT
* Septic shock or hemodynamic instability
* Stage 4 or greater chronic kidney disease
* Liver disease
* Decompensated heart failure
* Positive drug screen
* Receiving chemotherapy
* Immunocompromised
* Treatment with antiviral medication within 2 weeks prior to randomization
* Currently participating in another clinical trial
* Known phage allergy
* Pregnant/ breast feeding
* Lack of capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of phage + DAIR compared with placebo + DAIR in adult subjects with chronic or recalcitrant PJI | Day 1 through Week 24
  Incidence of reactions to study treatment and discontinuation due to adverse events
To evaluate the efficacy of phage + DAIR compared with placebo + DAIR in adult subjects with chronic or recalcitrant PJI | Day 1 through 24 months
  Time to recurrence or evidence of infection with the original pathogen at the same joint

SECONDARY OUTCOMES:
Treatment success | Day 1 through 12 months
  No recurrence or evidence of infection with the original pathogen at the same joint
No recurrence or evidence of infection for any reason | 12 months after DAIR
  Infection due to the original pathogen or a different pathogen

CONTACTS AND LOCATIONS:
Overall Officials: Edward Fang, MD, Study Chair — Adaptive Phage Therapeutics, Chief Medical Officer
Locations (10):
- United States (10):
  - University of California San Diego Medical Center, San Diego, California
  - Hartford Health Care Bone & Joint Insitute, Hartford, Connecticut
  - Snake River Research, Idaho Falls, Idaho
  - University of Maryland Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - New England Baptist Hospital, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - WVU Medicine JW Ruby Memorial Hospital, Morgantown, West Virginia